CLINICAL TRIAL: NCT01331070
Title: Central Control of Breathing in Patients With Chronic Obstructive Pulmonary Disease: Identification and Dynamics With Cerebral Functional Magnetic Resonance Imaging
Brief Title: Identification and Dynamics With Cerebral Functional Magnetic Resonance Imaging
Acronym: CHAOSBOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P100136; AOM10010 (Other: French Ministry)
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PATIENT (Experimental): Patients, half with moderate (GOLD II) and half with severe (GOLD III) COPD
  Interventions: Other: cerebral fMRI
- Accepts Healthy Volunteers (Other): Control arm with the same intervention
  Interventions: Other: cerebral fMRI

INTERVENTIONS:
Other: cerebral fMRI — the central breathing control with cerebral fMRI in COPD patients
  Other Names: the central breathing control with cerebral fMRI
  Arms: PATIENT
Other: cerebral fMRI — the central breathing control with cerebral fMRI in Accepts Healthy Volunteers
  Other Names: the central breathing control with cerebral fMRI
  Arms: Accepts Healthy Volunteers

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronicle inflammatory disease with a non reversible diminution of the airway flow. COPD is caused most commonly from tobacco smoking, which triggers an abnormal inflammatory response in the lung. Worldwide, COPD ranked as the sixth leading cause of death in 1990. It is projected to be the fourth leading cause of death worldwide by 2030 due to an increase in smoking rates and demographic changes in many countries. COPD is responsible for 16000 deaths per year in France, 100 000 hospitalizations per year and the health care expenditure of COPD in France is 3.5 billion of Euros. Classical markers of the disease severity, the forced expiratory volume in one second, poorly correlates with dyspnea and prognosis. Therefore, many studies focused on the control of breathing in an attempt to understand the pathophysiological mechanisms involved in the progression of the disease. Breathing control is enhanced in patients with COPD due to the progressive failure of respiratory muscles (airflow obstruction, static and dynamic hyperinflation, positive intrinsic end expiratory pressure), the ventilation/ perfusion ratio abnormalities leading to the loss of the gaz exchange efficiency. Inspiratory command depends on the medulla automatic pathway and the voluntary corticospinal command. Indirect method of breathing control estimation suggested in COPD patients an increased excitability of neurons involved in the voluntary diaphragm activation and a reduced cortical reserve. This may represent an increase risk factor for acute respiratory failure. Until now, no study reported the central breathing control with cerebral fMRI in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a chronicle inflammatory disease with a non reversible diminution of the airway flow. COPD is caused most commonly from tobacco smoking, which triggers an abnormal inflammatory response in the lung. Worldwide, COPD ranked as the sixth leading cause of death in 1990. It is projected to be the fourth leading cause of death worldwide by 2030 due to an increase in smoking rates and demographic changes in many countries. COPD is responsible for 16000 deaths per year in France, 100 000 hospitalizations per year and the health care expenditure of COPD in France is 3.5 billion of Euros. Classical markers of the disease severity, the forced expiratory volume in one second, poorly correlates with dyspnea and prognosis. Therefore, many studies focused on the control of breathing in an attempt to understand the pathophysiological mechanisms involved in the progression of the disease. Breathing control is enhanced in patients with COPD due to the progressive failure of respiratory muscles (airflow obstruction, static and dynamic hyperinflation, positive intrinsic end expiratory pressure), the ventilation/ perfusion ratio abnormalities leading to the loss of the gaz exchange efficiency. Inspiratory command depends on the medulla automatic pathway and the voluntary corticospinal command. Indirect method of breathing control estimation suggested in COPD patients an increased excitability of neurons involved in the voluntary diaphragm activation and a reduced cortical reserve. This may represent an increase risk factor for acute respiratory failure. Until now, no study reported the central breathing control with cerebral fMRI in COPD patients. This pilot study also aims in estimating if the absence or diminution of the cortical reserve is a marker of disease severity. In addition correlations will be performed between activated neuronal signals with fMRI and ventilatory flow output recordings (chaotic analysis).

ELIGIBILITY:
INCLUSION CRITERIA for Patient:

* Informed patients with written consent,
* More than eighteen years old,
* Patients having a social insurance
* A previous medical examination
* Patients, half with moderate (GOLD II) and half with severe (GOLD III) COPD will be included. These patients will be clinically in a steady state situation for at least one month (no acute exacerbation). GOLD grading of COPD patients will be performed according to the American Thoracic Society.

EXCLUSION CRITERIA for patient:

* Long-term oxygen therapy
* Previous cerebral vascular accident
* Central neurological disease (tumor, Parkinson, etc.)
* Nobody benefiting from a particular protection: pregnant woman, minor person, major person under guardianship and under guardianship, the persons hospitalized without their consent and protected by the law, or the private persons of freedom.
* Contraindication in the functional intellectual MRI:
* Port of a biomedical device like cardiac simulator
* Cardiac defibrillator
* Insulin pump or neurostimulating,
* Claustrophobia,
* Impossibility to remain lengthened
* Presence of cerebral vascular clips, metallic foreign body intra-ocular, not compatible cardiac valve
* Pregnancy

INCLUSION CRITERIA for Healthy Volunteers:

* Informed healthy volunteer with written consent,
* More than eighteen years old,
* Healthy volunteer having a social insurance
* A previous medical examination
* Non-smoker
* Non pathology and medicinal treatment

EXCLUSION CRITERIA for healthy volunteers:

* Nobody benefiting from a particular protection: pregnant woman, minor person, major person under guardianship and under guardianship, the persons hospitalized without their consent and protected by the law, or the private persons of freedom.
* Contraindication in the functional intellectual MRI:
* Port of a biomedical device like cardiac simulator
* Cardiac defibrillator
* Insulin pump or neurostimulating,
* Claustrophobia,
* Impossibility to remain lengthened
* Presence of cerebral vascular clips, metallic foreign body intra-ocular, not compatible cardiac valve
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Central ventilatory control | 1 month
  Evaluation of the central ventilatory control at the patients COPD during the application of an inspiratory resistance.

SECONDARY OUTCOMES:
Evaluation of the neuronal activation | 1 month
  Evaluation of the neuronal activation bulbo-pontique and corticospinal during the application of an inspiratory resistance.
Chaotic analysis | 1 month
  The correlations will be performed between activated neuronal signals with fMRI and ventilatory flow output recordings (chaotic analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Laurence MANGIN, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France